CLINICAL TRIAL: NCT00688350
Title: Interventions to Improve Medication-Taking Behavior in Older Adults With Hypertension: An Exploratory Study
Brief Title: Medication Adherence in Hypertension Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: The John A. Hartford Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMC1114797
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
Keywords: Hypertension; Aging; Medication adherence; Medication compliance
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral feedback (Experimental): Behavioral feedback intervention to improve adherence to antihypertensive medication
  Interventions: Behavioral: Behavioral feedback
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Behavioral feedback — The medication adherence intervention consists of five components: medication feedback, hypertension feedback, medication-taking skills, habit adjustment, and succinct medication and disease information delivered over an 8-week period.
  Arms: Behavioral feedback

SUMMARY:
The purpose of this study is to test an intervention to help older adults do a better job of following blood pressure medication regimens prescribed by their health care providers.

DETAILED DESCRIPTION:
Hypertension is present in 26.7% of the U.S. adult population between ages 20 to 74 (National Center for Health Statistics, 2006). The prevalence increases with age. Sixty-seven percent of adults aged 60 years or older have hypertension, a rise from 58% just ten years earlier (Ostchega, Dillon, Hughes, Carroll, & Yoon, 2007). Uncontrolled hypertension increases the risk for heart attack, stroke, congestive heart failure, and kidney disease (Chobanian et al., 2003; Stamler, Stamler, & Neaton, 1993; Vasan et al., 2001). Maintaining a normal blood pressure has been shown to be associated with a greater probability of living to age 85, and of living to age 85 without major health concerns (Terry et al., 2005). The most common treatment for managing hypertension involves the use of antihypertensive medications. These medications have been shown to effectively lower blood pressure (BP) and prevent the development of serious sequelae (Chobanian et al., 2003). Unfortunately, failure to adhere to antihypertensive medication regimens can impede the effectiveness of therapy.

Studies have reported levels of medication adherence among the elderly ranging from 26% to 59% (Botelho & Dudrak, 1992; van Eijken, Tsang, Wensing, de Smet, & Grol, 2003). Adherence to a medication regimen requires a set of behaviors that include obtaining the medication; timely administration of the correct drug, dose, and route; and persisting with taking the medication as long as the medication is needed. Success at these behaviors can be hampered by many of the changes often seen with age. Sensory loss, disturbances in memory and cognition, depression, and lifestyle changes such as retirement can disrupt routines or affect skills previously used to maintain medication adherence (Brown et al., 2005; Conn, Taylor, & Miller, 1994; Coons et al., 1994; Gehi, Haas, Pipkin, & Whooley, 2005; Schlenk, Dunbar-Jacob, & Engberg, 2004; Vik, Maxwell, & Hogan, 2004). Effective community-based interventions are needed to equip health care providers with tools to improve antihypertensive medication regimen adherence among their older patients. Many interventions have been tested to improve medication adherence in hypertension, but few addressing the unique needs of older adults. Of those that have been tested, there has been great variation in outcomes and ability to translate interventions into clinical practice.

This exploratory randomized controlled trial will test an 8-week behavioral intervention to improve medication adherence in older adults with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be aged 60 years or greater at time of study entry.
* Participants must be able to read, write, and converse in English.
* Participants will have a diagnosis of hypertension (based on participant report).
* Participants will have an active prescription for at least one antihypertensive medication with no antihypertensive prescription changes for 30 days at the time of study entry.
* Participants must self-administer his or her own medications without prompts from any other person or device.
* Baseline medication adherence rate of < 85%.
* Participants must be free of cognitive deficit as determined by a score of "normal" (0 - 2) on the Short Portable Mental Status Questionnaire (SPMSQ).
* Participants agree to complete all study contacts and measurements, including the use a special medication bottle with a Medication Event Monitoring System (MEMS) cap for the duration of the study.
* Able to open and close MEMS caps.

Exclusion Criteria:

* Participant is in state of severe hypertension (BP of >180/120 mmHg) at the time of study enrollment. Participants presenting with severely elevated blood pressure will be referred to their primary care provider.
* Participant resides in a residential facility where medications are administered by facility staff. Participants who reside in assisted living facilities but maintain control of their medications remain eligible.
* Participant has a terminal chronic illness with a life expectancy of six months or less.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: Medication adherence | 4 and 12 weeks post-intervention

SECONDARY OUTCOMES:
Resting blood pressure | 4 and 12 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Ruppar, PhD, RN, Principal Investigator — University of Missouri - Columbia Sinclair School of Nursing
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No